CLINICAL TRIAL: NCT06677151
Title: NPA-OSA Device Tolerability, Usability and Acclimation Clinical Study in Continuous Positive Airway Pressure (CPAP) Resistant Adult OSA Patients
Brief Title: NPA-OSA Device Tolerability, Usability and Acclimation Clinical Study in Adult Obstructive Sleep Apnea (OSA) Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Wallace H Coulter Center for Translational Research (Other)
Responsible Party: Principal Investigator, Louise O'Brien, Professor, Sleep Medicine, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00179497
Record Dates: First submitted 2024-11-04; First posted 2024-11-06 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Sleep Apnea, Obstructive
Keywords: nasopharyngeal
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Nasopharyngeal airway device (Experimental): A nasopharyngeal airway obstructive sleep apnea ("NPA"-OSA) device will be used for one night in a sleep laboratory and 30 days at home.
  Interventions: Device: nasopharyngeal airway obstructive sleep apnea (NPA-OSA) device

INTERVENTIONS:
Device: nasopharyngeal airway obstructive sleep apnea (NPA-OSA) device — The NPA-OSA is a flexible, medical-grade silicone, tube-like device that is self-inserted into the user's nasopharyngeal airway through one nostril prior to sleep and worn throughout the night to reduce or alleviate snoring and obstructive sleep apnea.

SUMMARY:
This pilot study is being done to determine if the nasopharyngeal airway obstructive sleep apnea (NPA-OSA) device can be used in the treatment of OSA in adults. The researchers think that the NPA-OSA device will reduce the number of apneas.

ELIGIBILITY:
Inclusion Criteria:

* Capacity and willingness to sign consent
* Patient willingness to commit to and complete study over a 30-day time period
* Confirmed diagnosis of moderate to severe OSA (AHI >= 15)
* OSA caused by upper airway obstruction
* CPAP non-compliant where CPAP compliance is defined as using CPAP for at least 4 hours a night for at least 70% of nights or interest in an alternative sleep apnea therapy
* Adequate manual dexterity to demonstrate ability to self-insert and remove device

Exclusion Criteria:

* Within 3 months of initiating CPAP use, and actively using CPAP
* Supraglottic airway collapse
* Distal airway stenosis
* Tracheobronchomalacia
* Currently pregnant
* Active COVID-19 infection
* Need for anticoagulative therapy
* Severe nasal allergies
* Bleeding disorder
* More than mild elevation of End-tidal carbon dioxide (ETCO2) or total carbon dioxide (TCO2) values >60 mmHg for >10% of sleep time
* Restrictive thoracic disorders
* Silicone, lidocaine, neosynephrine allergy
* Recurrent epistaxis
* Uncontrolled or serious illness, included but not limited to: severe breathing disorders including hypercapnic respiratory failure, respiratory muscle weakness, bullous lung disease (as seen in some types of emphysema), bypassed upper airway, pneumothorax, pneumomediastinum, etc.; severe heart disease (including heart failure); or pathologically low blood pressure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-07 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change in severity of apnea hypopnea index (AHI) | Baseline (day 0), 30 days
  The AHI is calculated by dividing the number of apnea events by the number of hours of sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Louise M O'Brien, PhD, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - Michigan Medicine, Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No